CLINICAL TRIAL: NCT00000640
Title: A Phase III Comparative Study of Dapsone / Trimethoprim and Clindamycin / Primaquine Versus Trimethoprim / Sulfamethoxazole in the Treatment of Mild-to-Moderate PCP in Patients With AIDS
Brief Title: A Phase III Comparative Study of Dapsone / Trimethoprim and Clindamycin / Primaquine Versus Sulfamethoxazole / Trimethoprim in the Treatment of Mild-to-Moderate PCP in Patients With AIDS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Jacobus Pharmaceutical (Industry); Glaxo Wellcome (Industry)
Responsible Party: Sponsor
Masking: Double | Purpose: Treatment
Other Study IDs: ACTG 108; 11083 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Pneumonia, Pneumocystis Carinii; HIV Infections
Keywords: Trimethoprim-Sulfamethoxazole Combination; Pneumonia, Pneumocystis carinii; Primaquine; Dapsone; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; Clindamycin; Sulfamethoxazole-Trimethoprim
MeSH Terms: conditions — Pneumonia, Pneumocystis; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Primaquine; Trimethoprim, Sulfamethoxazole Drug Combination; Dapsone; Clindamycin

INTERVENTIONS:
Drug: Primaquine
Drug: Sulfamethoxazole-Trimethoprim
Drug: Dapsone
Drug: Clindamycin

SUMMARY:
To evaluate the effectiveness of two oral treatments for mild to moderate Pneumocystis carinii pneumonia (PCP): dapsone/trimethoprim or clindamycin/primaquine as compared to a standard treatment program of sulfamethoxazole/trimethoprim (SMX/TMP) to assess the tolerance of these two alternative treatments as compared to the standard treatment of SMX/TMP. Per 09/09/92 amendment, to assess the efficacy and tolerance of these two alternative treatments in patients who are intolerant to SMX/TMP.

The type of treatment being studied has the advantages of wide applicability throughout the world (including developing countries) and low cost. An oral treatment is more accessible to patients than drugs given by injection or by inhalation.

DETAILED DESCRIPTION:
The type of treatment being studied has the advantages of wide applicability throughout the world (including developing countries) and low cost. An oral treatment is more accessible to patients than drugs given by injection or by inhalation.

Patients with confirmed PCP are randomized into one of three treatment groups. Group A receives SMX/TMP. Half of group A receives dapsone placebo (placebo is an inactive substance) daily plus trimethoprim placebo; the other half receives clindamycin placebo plus primaquine placebo. Group B is given dapsone plus trimethoprim. Half of group B receives SMX/TMP placebo; the other half receives clindamycin placebo plus primaquine placebo. Group C is given clindamycin plus primaquine. Half of group C receives SMX/TMP placebo, the other half receives dapsone placebo plus trimethoprim placebo. Treatment lasts 21 days; dosages will be adjusted for patients weighing less than 50 kg and more than 80 kg. Patients with a history of intolerance to SMX/TMP for whom rechallenge is considered medically contraindicated may be randomized to one of the non-sulfamethoxazole-containing arms.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Erythropoietin.
* Maintenance treatment with investigational triazoles (e.g., itraconazole).
* Antiemetics for nausea/vomiting, antihistamines for rash/pruritus, antipyretics for systemic symptoms (fever, headache, etc.) should be used for treatment of symptoms.
* Nonsteroidal antiinflammatory agents may be used for control of myalgias, headache, etc.

Concurrent Treatment:

Allowed:

* Blood transfusions.

Patients must have the following:

* Pneumocystis carinii pneumonia.
* HIV infection.
* Willing and able to sign informed consent. Patients under 18 years of age may enter with consent of parent or guardian.

Prior Medication:

Allowed:

* Up to 24 hours of treatment with sulfamethoxazole/trimethoprim (SMX/TMP), dapsone / trimethoprim, or clindamycin / primaquine, or one dose of pentamidine for this episode of Pneumocystis carinii pneumonia (PCP).
* Prior PCP prophylaxis.

Required:

* Adjunctive prednisone therapy in patients with (A-a) DO2 of 35 - 45 torr receiving acute anti-PCP treatment.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions and diseases are excluded:

Positive screen for glucose-6-phosphate dehydrogenase deficiency.

* Known NAD methemoglobin reductase deficiency and/or known hemoglobin M abnormality.

Concurrent Medication:

Excluded:

* Zidovudine (AZT).
* Ganciclovir.
* GM-CSF or G-CSF. Rifampin.
* Rifabutin.
* Corticosteroids (in patients with baseline (A-a) DO2 < 35 torr). Investigational drugs not specifically allowed.
* Folinic acid.

Patients with the following are excluded:

* Previous dose-limiting intolerance to sulfones, trimethoprim, clindamycin, or primaquine.

Requirement for other medications potentially effective in the treatment of Pneumocystis carinii pneumonia (PCP) (e.g., pyrimethamine and sulfadiazine).

* Prior enrollment in ACTG 108. Presence of other concurrent pulmonary pathology that would make interpretation of response to antipneumocystis therapy difficult.

Inability to take oral therapy.

Prior Medication:

Excluded:

* Acute treatment doses of anti-Pneumocystis carinii pneumonia agents within 30 days prior to study entry except as noted above.
* Systemic steroids above adrenal replacement doses within 7 days prior to study entry (except for patients with (A-a) DO2 of 35 - 45 torr who receive prednisone in conjunction with acute anti-PCP treatment).

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 290
Dates: Study Completion 1994-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Safrin S, Study Chair; Black JR, Study Chair
Locations (32):
- United States (32):
  - USC CRS, Los Angeles, California
  - Stanford CRS, Palo Alto, California
  - Ucsf Aids Crs, San Francisco, California
  - Santa Clara Valley Med. Ctr., San Jose, California
  - San Mateo County AIDS Program, San Mateo, California
  - Harbor-UCLA Med. Ctr. CRS, Torrance, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Univ. of Hawaii at Manoa, Leahi Hosp., Honolulu, Hawaii
  - Rush Univ. Med. Ctr. ACTG CRS, Chicago, Illinois
  - Northwestern University CRS, Chicago, Illinois
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - Methodist Hosp. of Indiana, Indianapolis, Indiana
  - Tulane Med. Ctr. - Charity Hosp. of New Orleans, ACTU, New Orleans, Louisiana
  - Johns Hopkins Adult AIDS CRS, Baltimore, Maryland
  - Massachusetts General Hospital ACTG CRS, Boston, Massachusetts
  - Beth Israel Deaconess - East Campus A0102 CRS, Boston, Massachusetts
  - University of Minnesota, ACTU, Minneapolis, Minnesota
  - Washington U CRS, St Louis, Missouri
  - SUNY - Buffalo, Erie County Medical Ctr., Buffalo, New York
  - Beth Israel Med. Ctr. (Mt. Sinai), New York, New York
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Cornell University A2201, New York, New York
  - NYU Med. Ctr., Dept. of Medicine, New York, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - Unc Aids Crs, Chapel Hill, North Carolina
  - Carolinas HealthCare System, Carolinas Med. Ctr., Charlotte, North Carolina
  - Regional Center for Infectious Disease, Wendover Medical Center CRS, Greensboro, North Carolina
  - Univ. of Cincinnati CRS, Cincinnati, Ohio
  - Case CRS, Cleveland, Ohio
  - The Ohio State Univ. AIDS CRS, Columbus, Ohio
  - Pitt CRS, Pittsburgh, Pennsylvania
  - University of Washington AIDS CRS, Seattle, Washington

REFERENCES:
- [Background] Wu AW, Gray S, Brookmeyer R, Safrin S. Quality of life in a double-blind randomized trial of 3 oral regimens for mild-to-moderate Pneumocystis carinii pneumonia in AIDS (ACTG 108). Int Conf AIDS. 1996 Jul 7-12;11(1):229 (abstract no TuB112)
- [Background] Safrin S, Finkelstein DM, Feinberg J, Frame P, Simpson G, Wu A, Cheung T, Soeiro R, Hojczyk P, Black JR. Comparison of three regimens for treatment of mild to moderate Pneumocystis carinii pneumonia in patients with AIDS. A double-blind, randomized, trial of oral trimethoprim-sulfamethoxazole, dapsone-trimethoprim, and clindamycin-primaquine. ACTG 108 Study Group. Ann Intern Med. 1996 May 1;124(9):792-802. doi: 10.7326/0003-4819-124-9-199605010-00003. PMID 8610948
- [Background] Rubin HR, Wu AW, Gutierrez M, Liriano O, Safrin S. Spanish translation of a functional status questionnaire for Pneumocystis carinii pneumonia. Int Conf AIDS. 1992 Jul 19-24;8(2):B178 (abstract no PoB 3549)